CLINICAL TRIAL: NCT05966649
Title: Synbiotics in Patients at RIsk fOr Preterm Birth: a Multi-center Double-blind Randomized Placebo-controlled trIal
Brief Title: Synbiotics in Patients at RIsk fOr Preterm Birth
Acronym: PRIORI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Z-2022080
Record Dates: First submitted 2023-03-02; First posted 2023-07-28 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-06

CONDITIONS: Preterm Spontaneous Labor With Preterm Delivery; Preterm Birth; Microbial Colonization
Keywords: Preterm birth; Vaginal microbiome; Probiotics; Synbiotics
MeSH Terms: conditions — Premature Birth; Communicable Diseases | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotics (Experimental): Oral synbiotic (food supplement) containing 8 probiotic Lactobacillus strains, the prebiotics inulin, fructooligosaccharides (FOS) and D-mannose.
  Interventions: Other: Synbiotics
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Synbiotics — Oral synbiotic (food supplement) containing 8 probiotic Lactobacillus strains, the prebiotics inulin, fructooligosaccharides (FOS) and D-mannose.
  Arms: Synbiotics
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Prematurity remains the main cause of death and serious health problems in new-borns. Besides the need for hospitalization and medical interventions in the first weeks or months of the new-borns' life, prematurity can cause long-lasting health problems (e.g. multiple hospital admissions, developmental delay, learning difficulties, motor delay, hearing or eye problems, ...). Moreover, prematurity places an enormous economic burden on the society. Aside from the medical problems and the financial cost, the emotional stress and psychological impact on the parents, siblings and other family members should not be underestimated.

Previous preterm delivery (before 37 weeks of pregnancy) increases the risk for recurrent preterm delivery in a subsequent pregnancy. Therefore, these women should be considered as 'high risk' for preterm birth.

Infections ascending from the vagina may be an important cause of preterm delivery in certain cases. Some women have an abnormal vaginal microbiome and are therefore at risk for infections and preterm birth. On the other hand, the vaginal flora is more stable and resistant to infections in healthy pregnant women who deliver at term (after 37 weeks of gestation).

Synbiotics are a mixture containing probiotics and prebiotics. Probiotics are living bacteria with potential beneficial effects that can be used safely in pregnancy, while prebiotics are consumed by the bacteria. It is known that probiotics, when used for a long period of time, can maintain a healthy and stable vaginal flora that may protect against infections. In this study, pregnant patients with a history of preterm birth will be included in the first trimester of pregnancy to start with synbiotics or placebo. The investigators will examine the effect of synbiotics on the vaginal flora and on the pregnancy duration. The hypothesis is that synbiotics, when started early in the pregnancy, can change the disturbed vaginal flora into a stable micro-environment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent must be obtained before any study assessment is performed;
2. 18 years of age or older;
3. Singleton pregnancy;
4. Pregnancy consultation between 8 and 10 weeks gestation.
5. At least one of the following risk factors for spontaneous preterm birth:

   * Prior spontaneous preterm birth, defined as delivery between 24 and 36 weeks following PPROM, preterm labor or cervical insufficiency
   * PPROM ≤36 weeks in previous pregnancy
   * Prior spontaneous second-trimester pregnancy loss, defined as PPROM, preterm labor or cervical insufficiency with birth between 14 and 24 weeks.

Exclusion Criteria:

1. Patients who are already using pro-, pre- or synbiotics and not willing to stop
2. Multiple pregnancy
3. Need for primary (type 1) cerclage
4. Inflammatory bowel disease
5. Known congenital uterine anomaly
6. History of LLETZ conization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery | Through study completion - at delivery

SECONDARY OUTCOMES:
Incidence of PTB, defined as GA at delivery < 37 weeks | Through study completion - at delivery
Proportion of PTB in different categories | Through study completion - at delivery
  * of patients that deliver < 28 weeks: extreme PTB
  * of patients that deliver from 28 until 37 weeks: very PTB
  * of patients that deliver from 32 until 37 weeks: moderate to late PTB
PPROM | Up to 34 weeks from the date of randomization
  Incidence
PPROM | Up to 34 weeks from the date of randomization
  Gestational age at PPROM
PPROM | Up to 34 weeks from the date of randomization
  Time to delivery
Composition of the vaginal microbiome | Assessed 3 times during the study period: at randomization, 11-13 weeks after randomization (at gestational age 19-21 weeks), and 21-23 weeks after randomization (29-31 weeks of gestation)
  The vaginal microbiome will be assessed throughout pregnancy at 4 well-defined stages of pregnancy (9, 20, 30 weeks and at delivery) and at admission at the MIC unit for preterm labor, PPROM or cervical insufficiency.
Incidence of neonatal admissions | Neonatal admission at a neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
Duration of neonatal admissions | Neonatal admission at a neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
Incidence of maternal admissions | Up to 34 weeks from the date of randomization
Duration of maternal admissions | Up to 34 weeks from the date of randomization
Quality Of Life during pregnancy and during neonatal admission at a neonatal intensive care unit | Trough study completion, on average 1 year
  Using EQ5D questionnaire (5 questions and scale from 1 to 100)
Neonatal outcome: infectious parameters | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Sepsis (early, late and culture negative), number of episodes (min 72 hours) of antibiotic treatment, duration of antibiotic treatment in days
Neonatal outcome: bronchopulmonary dysplasia (BPD) | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Proportion of each category (no, mild, moderate and severe)
Neonatal outcome: intraventricular haemorrhage | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Incidence
Neonatal outcome: periventricular leukomalacia | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Incidence
Neonatal outcome: respiratory support | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Need for respiratory support (CPAP: continuous positive airways pressure, non-invasive positive pressure ventilation or mechanical endotracheal ventilation) and the duration of respiratory support in days. Use and administration of surfactant
Neonatal outcome: retinopathy | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Incidence
Neonatal outcome: neonatal morbidity | During the admission at the neonatal intensive care unit (when the neonate is admitted at a neonatal intensive care unit within 7 days of delivery)
  Incidence
Neonatal outcome: birth weight | After the neonate is born

OTHER OUTCOMES:
Effect of antibiotics on the vaginal microbiome | During pregnancy until 28 days after PPROM
  When the patient is admitted in case the pregnancy was complicated with PPROM
Effect on the gastrointestinal microbiome of the neonate in case of PPROM | Between 13 to 36 weeks from the date of randomization
  When the neonate is born after a pregnancy complicated with PPROM
Placental microbiome in case of preterm birth | Between 13 to 36 weeks from the date of randomization
  In case the pregnancy was complicated with preterm birth (delivery before 37 weeks of gestation)

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (7):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Universitaire Ziekenhuizen Leuven, Leuven, Limburg
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - AZ Sint-Lucas, Bruges, West-Vlaanderen
  - AZ Groeninge, Kortrijk
  - CHR Citadelle, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nulens K, Papy E, Tartaglia K, Dehaene I, Logghe H, Van Keirsbilck J, Chantraine F, Masson V, Simoens E, Gysemans W, Bruckers L, Lebeer S, Allonsius CN, Oerlemans E, Steensels D, Reynders M, Timmerman D, Devlieger R, Van Holsbeke C. Synbiotics in patients at risk for spontaneous preterm birth: protocol for a multi-centre, double-blind, randomised placebo-controlled trial (PRIORI). Trials. 2024 Sep 17;25(1):615. doi: 10.1186/s13063-024-08444-8. PMID 39289685